CLINICAL TRIAL: NCT04216095
Title: Comparative Effectiveness Clinical Trial of Magnetic Seizure Therapy (MST) Compared to Electroconvulsive Therapy (MST) in Major Depressive Disorder
Brief Title: Comparative Effectiveness Clinical Trial of MST Compared to ECT in Major Depressive Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Nagy A. Youssef (Consultant on the MST technique) (Unknown)
Responsible Party: Principal Investigator, El-Sayed Gad, Professor, Tanta University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 025
Record Dates: First submitted 2019-12-23; First posted 2020-01-02 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Major Depressive Disorder
Keywords: MST; ECT; MDD; Depression; Major Depressive Disorder; Magnetic seizure therapy; Electroconvulsive Therapy; Treatment Resistant Depression (TRD)
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: MST (Magstim Theta device, Magstim Company Limited, Whitfield, Wales, UK) versus ECT (Thymatron IV device, Somatics LLC, USA) assigned per the clinical decision making of the ECT psychiatrist as deemed best for the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroconvulsive Therapy (ECT) (Active Comparator): Right unilateral (RUL, N=15), or Bitemporal (BT, N=15) ECT
  Interventions: Device: Electroconvulsive Therapy (n=30)
- Magnetic Seizure Therapy (MST) (Active Comparator): High-dose magnetic seizure therapy (HD-MST)
  Interventions: Device: Magnetic Seizure Therapy (n=30)

INTERVENTIONS:
Device: Electroconvulsive Therapy (n=30) — Right unilateral (RUL) ECT (n=15) or bitemporal (BT) ECT (n=15) using a Thymatron IV device (Somatics LLC, USA) twice weekly.
  Arms: Electroconvulsive Therapy (ECT)
Device: Magnetic Seizure Therapy (n=30) — High-dose magnetic seizure therapy (HD-MST) over the vertex using Magstim Theta device (Magstim Company Limited, Whitfield, Wales, UK) at 100% maximal output of the device (constant), with pulse frequency 100Hz and train duration 10 seconds twice weekly.
  Arms: Magnetic Seizure Therapy (MST)

SUMMARY:
This study was a prospective, open-label comparative effectiveness clinical trial, comparing magnetic seizure therapy (MST) to ECT in patients with Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
Magnetic seizure therapy (MST) has previously demonstrated fewer cognitive side effects than ECT in randomized trials of efficacy. However, there are currently no real-world effectiveness trials guided by the clinical decision making of the ECT psychiatrist as deemed best for the patient. The aims of this study are to: (1) Evaluate the comparative effectiveness of MST versus ECT in patients with MDD, and (2) Compare the cognitive adverse effects of MST and ECT, (3) Explore changes in SPECT that is associated with MST treatment and treatment response.

Patients will be clinically assigned to either ECT (n=30) or HD-MST (n=30) twice a week. Efficacy will be primarily assessed by the Hamilton Depression Rating Scale-21 (HAMD-21); primary cognitive side effects were assessed by Time to Reorientation (TRO) and secondarily cognitive battery. Brain SPECT will be done for patients before and after MST.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to consent
2. Clinically indicated for seizure therapy
3. Patients with MDD who had either never received antidepressant treatment or had discontinued antidepressants by their own choice for at least six weeks prior to enrollment (as commonly done in routine clinical care in this jurisdiction due to more negative views of psychotropics)
4. 18-65 years of age.

Exclusion Criteria:

1. Dementia,
2. Delirium
3. History of significant head trauma
4. Neurological disorders (e.g., epilepsy, stroke, multiple sclerosis)
5. Substance dependence
6. Active comorbidity with another psychiatric disorder
7. Patients who had previously received ECT or TMS
8. Current unstable or serious medical illness (e.g., myocardial infarction)
9. Pregnancy
10. Presence of implanted electronic devices (e.g., cardiac pacemaker, cochlear implants)
11. Inability to participate in testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06-07 (Actual); Primary Completion 2015-10-07 (Actual); Study Completion 2015-10-07 (Actual)

PRIMARY OUTCOMES:
Time to reorientation (TRO) | approximately 2.5 weeks
  Cognition primarily assessed by Time to Reorientation (TRO)
Depression Scale | approximately 2.5 weeks
  Efficacy primarily assessed by Hamilton Depression Scale-21 (HAM-D-21)

SECONDARY OUTCOMES:
Wechsler Memory Scale - Revised: | approximately 2.5 weeks
  Neuropsychological assessment
Wisconsin Card Sorting Test | approximately 2.5 weeks
  Neuropsychological assessment
Brain Single Photon Emission Computed Tomography (SPECT) | approximately 2.5 weeks
  Brain SPECT done for patients pre-post MST course to explore biological changes associated with MST and predictors of treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma El-Deeb, MD, PhD, Principal Investigator — Tanta University, Faculty of Medicine; El-Sayed Gad, MD, PhD, Principal Investigator — Tanta University, Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No